CLINICAL TRIAL: NCT02910518
Title: A Randomized, Double-blind, Single-dose, 2-Treatment, 2-Period, 2-Sequence Crossover Bioequivalence Study Comparing Two Formulations of Insulin Glulisine (Insulin Glulisine 300 Units/mL Versus Insulin Glulisine 100 Units/mL Marketed as Apidra® 100 Units/mL) Using the Euglycemic Clamp Technique, in Patients With Type 1 Diabetes Mellitus
Brief Title: A Study to Demonstrate Bioequivalence Between Insulin Glulisine U300 and Insulin Glulisine U100 After a Single Subcutaneous Dose Using the Euglycemic Clamp Technique, in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BEQ13941; 2016-001498-34 (EudraCT Number); U1111-1183-8636 (Other: UTN)
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — insulin glulisine; Insulin Aspart; Insulin, Isophane; Glucagon; Glucose; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin glulisine (U300) - Test formulation (Experimental): Insulin glulisine (U300) will be given as a single subcutaneous (SC) dose on Day 1 of each period under fasting conditions according to the random list and assigned sequence. Glucose, insulin aspart (IV) and heparin will be used for clamp procedure. NPH insulin (if necessary) and insulin aspart (SC) will be handed out at screening to change insulin regimen and glucagon at Day 1 to treat cases of severe hypoglycemia.
  Interventions: Drug: Insulin glulisine (U300); Drug: Insulin aspart; Drug: NPH insulin; Drug: Glucagon; Drug: Glucose; Drug: Heparin
- Insulin glulisine - Reference formulation (Active Comparator): Insulin glulisine (U100) will be given as a single SC dose on Day 1 of each period under fasting conditions according to the random list and assigned sequence. Glucose, insulin aspart (IV) and heparin will be used for clamp procedure. NPH insulin (if necessary) and insulin aspart (SC) will be handed out at screening to change insulin regimen and glucagon at Day 1 to treat cases of severe hypoglycemia.
  Interventions: Drug: Insulin glulisine; Drug: Insulin aspart; Drug: NPH insulin; Drug: Glucagon; Drug: Glucose; Drug: Heparin

INTERVENTIONS:
Drug: Insulin glulisine (U300) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: HMR1964 (U300)
  Arms: Insulin glulisine (U300) - Test formulation
Drug: Insulin glulisine — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Apidra®
  Arms: Insulin glulisine - Reference formulation
Drug: Insulin aspart — Pharmaceutical form: solution
  Route of administration: intravenous/subcutaneous
  Other Names: NovoRapid®
Drug: NPH insulin — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Insuman® Basal Solostar®
Drug: Glucagon — Pharmaceutical form: Powder and solvent for solution for injection
  Route of administration: subcutaneous
  Other Names: GlucaGen® HypoKit
Drug: Glucose — Pharmaceutical form: solution
  Route of administration: intravenous
  Other Names: Glucose 20%
Drug: Heparin — Pharmaceutical form: solution
  Route of administration: intravenous
  Other Names: Heparin-Natrium-5000

SUMMARY:
Primary Objective:

To demonstrate bioequivalence between insulin glulisine given as 300 Units/mL test formulation and insulin glulisine 100 Units/mL reference formulation after a single subcutaneous (SC) dose.

Secondary Objectives:

* To assess the pharmacodynamic (PD) profiles and further pharmacokinetic (PK) characteristics of insulin glulisine U300 in comparison to insulin glulisine U100 after a single SC dose.
* To assess safety and tolerability of the test and the reference formulation of insulin glulisine.

DETAILED DESCRIPTION:
The study duration per patient will be 18 to 62 days and will consist of a 4 to 28 days of screening period, a treatment period of 2 days, a washout between dosing occasions of 5-18 days, and follow up visit 7-14 days after last dosing.

ELIGIBILITY:
Inclusion criteria :

* Male or female subjects with type 1 diabetes mellitus (T1DM) for more than 1 year.
* Total insulin dose of <1.2 U/kg/day.
* Fasting negative serum C-peptide (<0.30 nmol/L).
* Glycohemoglobin at screening (HbA1c) ≤9%.
* Subjects with anti-insulin antibody titer at screening ≤30.0 kU/L.
* Stable insulin regimen for at least 2 months prior to study.
* Normal findings in medical history and physical examination (cardiovascular system, chest and lungs, thyroid, abdomen, nervous system, skin and mucosae, and musculoskeletal system), vital signs, electrocardiogram (ECG), and safety laboratory.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic (apart from T1DM), hematological, neurological, psychiatric, systemic (affecting the body as a whole), ocular, gynecologic (if female), or infectious disease; any acute infectious disease or signs of acute illness or any history or presence of heparin induced thrombocytopenia Type II (HIT-type II).
* Severe hypoglycemia resulting in coma/seizures or requiring assistance of another person, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Frequent severe headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).
* Symptomatic hypotension (whatever the decrease in blood pressure), or asymptomatic postural hypotension defined by a decrease in systolic blood pressure equal to or greater than 20 mmHg within three minutes when changing from the supine to the standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* Any medication (including medicine containing St John's Wort) within 14 days before inclusion (for systemic glucocorticoids within 3 months) or within 5 times the elimination half-life or PD half-life of the medication, with the exception of insulin, stable treatment (at least 2 months) with thyroid hormones, lipid-lowering and antihypertensive drugs and if female with the exception of hormonal contraception or menopausal hormone replacement therapy.
* Positive reaction to any of the following tests: hepatitis B surface (HBs Ag) antigen, anti hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Assessment of PK parameter: maximum observed insulin concentration | 10 hours
Assessment of PK parameter: area under the concentration time curve | 10 hours

SECONDARY OUTCOMES:
Assessment of PK parameter: time to reach Cmax (INS-tmax) | 10 hours
Assessment of PK parameter: terminal half-life (INS-t1/2z) | 10 hours
Assessment of PD parameter: area under the body weight standardized glucose infusion rate (GIR) versus time curve from 0 to 10 hours (GIR-AUC0-10) | 10 hours
Assessment of PD parameter: maximum smoothed body weight standardized GIR (GIRmax) | 10 hours
Assessment of PD parameter: time to GIRmax (GIR-tmax) | 10 hours
Duration of blood glucose control under clamp conditions - time | 10 hours
Number of patients with treatment emergent adverse events | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org